CLINICAL TRIAL: NCT04546633
Title: A Phase 2 Interventional, Multicenter, Randomized, Open-label Study in Three Age-descending Cohorts to Evaluate Efficacy, Safety and Tolerability of KAF156 and Lumefantrine-SDF Combination in the Treatment of Acute Uncomplicated Plasmodium Falciparum Malaria in a Pediatric Population
Brief Title: Efficacy, Safety and Tolerability of KAF156 in Combination With Lumefantrine Solid Dispersion Formulation (LUM-SDF) in Pediatric Population With Uncomplicated Plasmodium Falciparum Malaria
Acronym: KALUMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CKAF156A2203; 2021-003583-27 (EudraCT Number)
Record Dates: First submitted 2020-09-05; First posted 2020-09-14 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Uncomplicated Plasmodium Falciparum Malaria
Keywords: Plasmodium falciparum malaria; KAF156; Lumefantrine Solid Dispersion Formulation; LUM-SDF; children
MeSH Terms: conditions — Malaria, Falciparum | interventions — ganaplacide; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label, randomized study in adolescents and children with confirmed uncomplicated P. falciparum malaria.
  This study will first explore the effect of food on lumefantrine and KAF156 PK in a Run-in Cohort of patients 12 to < 18 years old with malaria caused by P. falciparum, before younger patients are assessed. Then, efficacy, safety and tolerability of the combination of KAF156 and LUM-SDF will be evaluated in younger patients, first in Cohort 1 of patients 2 to < 12 years old and then in Cohort 2 of patients 6 months to < 2 years old.
  Randomization is stratified by country for patients in the Run-in cohort, by age group (6 years to <12 and 2 to <6 years) and country in Cohort 1 and by country in Cohort 2.
Who Masked: Outcomes Assessor
Masking Description: Treatment and food condition during the Run-in cohort will be open to patients/patients' parents/legal guardian, investigators staff and study monitors, as well as to the Clinical Trial Team (CTT) to allow continuous review of safety, drug exposure and efficacy data in pediatric population. For Cohorts 1 and 2, treatment/food condition will be open to patients/patients' parents/legal guardian, investigators staff and study monitors but will be blinded to the Clinical Trial Team (CTT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Run-in - KAF156 and LUM-SDF QD for 2 days in fasted condition (Experimental): KAF156 and LUM-SDF QD (once daily) for 2 days in fasted condition
  Interventions: Drug: KAF156; Drug: LUM-SDF
- Run-in - KAF156 and LUM-SDF QD for 2 days in fed condition (Experimental): KAF156 and LUM-SDF QD (once daily) for 2 days in fed condition
  Interventions: Drug: KAF156; Drug: LUM-SDF
- Cohort 1/2 - KAF156 and LUM-SDF QD (once daily) in either a 2-day or 3-day dose regimen (Experimental): KAF156 and LUM-SDF QD (once daily) in either a 2-day or 3-day dose regimen. Food recommendation will be issued after the Run-in Cohort based on efficacy, safety, tolerability and PK data).
  Interventions: Drug: KAF156; Drug: LUM-SDF
- Cohort 1/2 - Coartem® BID (twice a day) for 3 days (Active Comparator): Coartem® BID (twice a day) for 3 days (will be administered with food and doses will be based on patient's body weight as per product label).
  Interventions: Drug: Coartem

INTERVENTIONS:
Drug: KAF156 — Provided as 50 mg or 100 mg tablets, to be taken QD 2 or 3 Days in combination with LUM-SDF, dose is based on body weight
  Arms: Cohort 1/2 - KAF156 and LUM-SDF QD (once daily) in either a 2-day or 3-day dose regimen; Run-in - KAF156 and LUM-SDF QD for 2 days in fasted condition; Run-in - KAF156 and LUM-SDF QD for 2 days in fed condition
Drug: LUM-SDF — Provided as 60 mg, 120 mg or 240 mg powder in sachet, to be taken QD 2 or 3 Days in combination with KAF156, dose is based on body weight
  Other Names: Lumefantrine Solid Dispersion Formulation
  Arms: Cohort 1/2 - KAF156 and LUM-SDF QD (once daily) in either a 2-day or 3-day dose regimen; Run-in - KAF156 and LUM-SDF QD for 2 days in fasted condition; Run-in - KAF156 and LUM-SDF QD for 2 days in fed condition
Drug: Coartem — Coartem® (dispersible tablets in blister pack) (for Cohorts 1 and 2), dose is based on body weight
  Arms: Cohort 1/2 - Coartem® BID (twice a day) for 3 days

SUMMARY:
This study aims to determine the efficacy, safety and tolerability of the investigational drug KAF156 in combination with a solid dispersion formulation of lumefantrine (LUM-SDF) in pediatric patients (6 months to < 18 years of age) with uncomplicated P. falciparum malaria. There is an unmet medical need for anti-malarial treatment with a new mechanism of action to reduce the probability of developing resistance.

DETAILED DESCRIPTION:
This Phase 2 study aims to evaluate the efficacy, safety and tolerability of the investigational drug KAF156 and a Solid Dispersion Formulation of lumefantrine (LUM-SDF) when administered in combination in pediatric patients 6 months to < 18 years of age with uncomplicated Plasmodium falciparum malaria. In addition, pharmacokinetics (PK) of the drug combination will also be evaluated.

There will be three age-descending cohorts: Run-in Cohort, Cohort 1 and Cohort 2.

It is important to understand the impact of food on exposure. In adult healthy volunteers, LUM-SDF alone has shown a food effect whereas KAF156 does not have a food effect. This new study will first explore the effect of food on lumefantrine and KAF156 PK in malaria patients 12 to < 18 years old with malaria caused by P. falciparum before younger patients are assessed.

Then, efficacy, safety and tolerability of the combination of KAF156 and LUM-SDF will be evaluated in younger patients, first in Cohort 1 of patients 2 to < 12 years old and then in Cohort 2 of patients 6 months to < 2 years old.

ELIGIBILITY:
Inclusion Criteria:

1. In run-in cohort: Male and female patients 12 to < 18 years of age, with a body weight

   * 35.0 kg In Cohort 1: Male and female patients 2 to < 12 years of age, with a body weight ≥ 10.0 kg In Cohort 2: Male and female patients 6 months to < 2 years of age, with a body weight
   * 5.0 kg
2. Microscopic confirmation of P. falciparum by Giemsa-stained thick and thin films
3. P. falciparum parasitemia of ≥ 1,000 and ≤ 150,000 parasites/μL at the time of prescreening for the Run-in Cohort; and P. falciparum parasitemia of ≥ 1,500 and ≤ 150,000 parasites/μL at the time of pre-screening for Cohorts 1 and 2
4. Axillary temperature ≥ 37.5 ºC or oral/tympanic/rectal temperature ≥ 38.0 ºC; or history of fever during the previous 24 hours (at least documented verbally)
5. Written informed consent has been obtained from parent / legal guardian before any assessment is performed. If the parent/legal guardian is unable to read and write, then a witnessed consent according to local ethical standards is permitted. Patients who are capable of providing assent, must provide assent with parental/legal guardian consent or as per local ethical guidelines
6. The patient and his/her parent/legal guardian is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions and is likely to complete the study as planned

Exclusion Criteria:

1. Mixed Plasmodium infections as per light microscopy results
2. Signs and symptoms of severe malaria according to WHO 2015 (see Section 16.4)
3. Significant, non-plasmodial co-infections including tuberculosis
4. Patients with concurrent febrile illnesses (e.g., typhoid fever, known or suspected COVID19)
5. Known relevant liver disease e.g. chronic hepatitis, cirrhosis, compensated or decompensated, history of hepatitis B or C, hepatitis B or A vaccination in last 3 months, known gallbladder or bile duct disease, acute or chronic pancreatitis
6. Major congenital defects
7. Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection or family history of congenital or hereditary immunodeficiency
8. Immunosuppressive therapy (steroids, immune modulators or immune suppressors) within 3 months prior to recruitment. (For corticosteroids, this will mean prednisone, or equivalent, ≥ 0.5 mg/kg/day. Inhaled and topical steroids are allowed)
9. Repeated vomiting (defined as more than 3 times in the 24 hours prior to inclusion in the study) or severe diarrhea (defined as more than 3 watery stools in the 24 hours prior to inclusion in the study)
10. Active duodenal ulcer, ulcerative colitis, Crohn's disease, chronic (i.e., > 2 weeks) use of non-steroidal anti-inflammatory drugs (NSAIDs)
11. Clinically relevant abnormalities of electrolyte balance which require correction, e.g., hypokalemia, hypocalcemia or hypomagnesemia
12. Anemia (hemoglobin level <7 g/dL)
13. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs (e.g., HIV patients on ART therapy or TB patients on treatment), or which may jeopardize the patient in case of participation in the study. The investigator should make this determination in consideration of the patient's medical history and/or clinical or laboratory evidence of any of the following:

    * AST/ALT > 3 x the upper limit of normal range (ULN), regardless of the level of total bilirubin
    * AST/ALT > 1.5 and ≤ 2 x ULN and total bilirubin is > ULN Total bilirubin > 2 x ULN regardless of the level of AST/ALT
14. Resting QT interval corrected by Fridericia's formula (QTcF) > 450 ms at screening
15. Creatinine > 2 x ULN in the absence of dehydration. In case of dehydration, creatinine should be < 2 x ULN after oral/parenteral rehydration
16. Any severe disease condition which might prohibit participation in this study
17. Known chronic underlying disease such as sickle cell disease, and severe cardiac, renal, or hepatic impairment
18. Known active or uncontrolled thyroid disease
19. Inability to swallow oral medication (in tablet and/or liquid form)
20. Patients with prior antimalarial therapy or antibiotics with antimalarial activity within minimum of their five (5) plasma half-lives (or within 4 weeks of screening if half-life is unknown)
21. Use of other investigational drugs within 30 days of dosing or until the expected pharmacodynamic effect has returned to baseline, whichever is longer
22. Patients taking medications prohibited by the protocol
23. Previous participation in any malaria vaccine study or received malaria vaccine in any other circumstance within 3 months of dosing
24. History or family history of long QT syndrome or sudden cardiac death, or any other clinical condition known to prolong the QTc interval, such as history of symptomatic cardiac arrhythmias, clinically relevant bradycardia or severe heart disease
25. Use of agents known to prolong the QT interval unless it can be permanently discontinued for the duration of study
26. History of hypersensitivity to any of the study drugs or its excipients or to drugs of similar chemical classes

    For the Run-in Cohort only:
27. Pregnant or nursing (lactating) patients
28. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception during dosing of investigational drug. Basic contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking investigational drug. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 m prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps).

    Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking investigational drug. Women are considered not of child bearing potential if they have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

    For Cohorts 1 and 2 only:
29. Patients of child bearing potential, defined as all girls post first menarche (except for Run-in Cohort)

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 295 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
PCR-corrected adequate clinical and parasitological response (ACPR) at Day 29 (i.e., 28 days post-dose) (Cohorts 1 and 2 pooled). | Day 29
  The primary efficacy variable is the PCR corrected Adequate Clinical and Parasitological Response (ACPR) at Day 29 (Cohorts 1 and 2 pooled). In case that Cohort 2 stops early, such as after the first 24 patients, the study objectives will be assessed based on Cohort 1 data alone. A patient is considered as PCR corrected ACPR at Day 29 if the patient does not meet any of the criteria of early treatment failure (ETF) (up to Day 4), late clinical failure (LCF) (Day 5 to Day 29) or late parasitological failure (LPF) (Day 8 to Day 29), and is absence of parasitaemia on Day 29 irrespective of axillary temperature unless the presence of parasitaemia after 7 days (Day 8 or later) is due to reinfection based on PCR genotyping. A presence of parasitaemia after 7 days of treatment initiation is considered as a reinfection only if the parasitaemia is clear before Day 8 and none of the parasite strain(s) detected on Day 8 or later match with the parasite strain at baseline based on PCR genotyping.

SECONDARY OUTCOMES:
Percentage of Participants with Polymerase Chain Reaction (PCR)-corrected and uncorrected Adequate Clinical and Parasitological Response (ACPR) at Day 15 and 43 | Day 15, Day 43
  A blood draw will be performed at each collection time point for parasitemia assessment.
Percentage of Participants with Polymerase Chain Reaction (PCR)-corrected and uncorrected Adequate Clinical and Parasitological Response (ACPR) at Day 29 (Run-in Cohort) | Day 29
  A blood draw will be performed at Day 29 in the Run-in Cohort only for parasitemia assessment.
Time to parasite clearance (PCT) | up to 43 days
  Parasite Clearance Time (PCT) is defined as the time from the first dose until the first total and continued disappearance of asexual parasite forms which remained at least a further 48 hours.
Time to fever clearance (FCT) | up to 43 days
  Fever Clearance Time (FCT) is defined as the time from the first dose until the first time the axillary body temperature decreased below and remained below 37.5°C axillary or 38.0°C oral/tympanic/rectal for at least a further 24 hours.
Proportion of patients with Early Treatment Failure (ETF) | Day 1 to Day 4
  ETF is defined as:
  * Development of danger signs or severe malaria on Day 2, Day 3, Day 4 in the presence of parasitemia
  * Parasitemia on Day 3 higher than Day 1 count irrespective of axillary temperature
  * Parasitemia on Day 4 with axillary temperature ≥ 37.5°C
  * Parasitemia on Day 4 equals to or more than 25% of count on Day 1
Proportion of patients with Late Clinical Failure (LCF) | Day 5 to Day 43
  LCF is defined as:
  * Development of danger signs or severe malaria on any day from Day 5 to Day 43 in the presence of parasitemia without previously meeting any of the criteria of ETF
  * Presence of parasitemia and axillary temperature ≥ 37.5oC on any day from Day 5 to Day 43 without previously meeting any of the criteria of ETF
Proportion of patients with Late Parasitological Failure (LPF) | Day 8 to Day 43
  LPF is defined as the presence of parasitemia on any day from Day 8 to Day 43 and axillary temperature < 37.5oC without previously meeting any of the criteria of ETF or LCF
Incidence rate of recrudescence and reinfection | Day 15, Day 29 and Day 43
  Time to event (recrudescence or reinfection) will be calculated from the time of first study medication to the date of first event if a patient experiences the event and be censored at the time of last parasite assessment if a patient does not experience the event due to whatever reason.
  Reinfection is defined as appearance of asexual parasites after clearance of initial infection with a genotype different from those parasites present at baseline.
  Recrudescence is defined as appearance of asexual parasites after clearance of initial infection with a genotype identical to that of parasites present at baseline.
  Reinfection and Recrudescence must be confirmed by PCR analysis.
Number of Participants with On-Treatments Adverse Events, Serious Adverse Events, and Deaths | Day 1 to Day 43
  Analysis of absolute and relative frequencies for treatment emergent Adverse Event (AE), Serious Adverse Event (SAE) and Deaths by primary System Organ Class (SOC) to demonstrate that KAF156 and Lumefantrine-SDF combination, under fasted or fed conditions is safe through the monitoring of relevant clinical and laboratory safety parameters.
Pharmacokinetics of KAF156 and LUM-SDF PK (Run-in Cohort, Cohort 1 and 2): Area Under the Plasma Concentration-time Curve (AUC) | From Day 1 to Day 8
  AUC is the area under the plasma concentration-time curve. PK parameters were calculated from plasma concentration-time data using non-compartmental methods.
Pharmacokinetic of KAF156 and LUM-SDF PK (Run-in Cohort, Cohort 1 and 2): Maximum Observed Plasma Concentration (Cmax) | From Day 1 to Day 8
  Cmax is the maximum observed plasma concentration following drug administration. PK parameters are calculated from plasma concentration-time data using non-compartmental methods.
Pharmacokinetic of KAF156 and LUM-SDF PK (Run-in Cohort, Cohort 1 and 2): Time to reach the maximum concentration after drug administration (Tmax) | From Day 1 to Day 8
  Tmax is the time to reach maximum plasma concentration following drug administration. PK parameters are calculated from plasma concentration-time data using non-compartmental methods.
Pharmacokinetics of KAF156 and LUM-SDF PK (Run-in Cohort, Cohort 1 and 2): Plasma drug concentration 168 hours post first dose administration (C168h) | Day 8
  C168h is the plasma concentration at 168h post first dose administration.
Pharmacokinetics of LUM from Coartem arm (Cohorts 1 and 2): Maximum Observed Plasma Concentration (Cmax) | From Day 1 to Day 8
  Cmax is the maximum observed plasma concentration following drug administration. PK parameters are calculated from plasma concentration-time data using non-compartmental methods.
Pharmacokinetics of LUM from Coartem arm (Cohorts 1 and 2): Plasma drug concentration 168 hours post first dose administration (C168h) | Day 8
  C168h is the plasma concentration at 168h post first dose administration.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Burkina Faso (4):
  - Novartis Investigative Site, Banfora
  - Novartis Investigative Site, Bobo-Dioulasso
  - Novartis Investigative Site, Ouagadougou
  - Novartis Investigative Site, Sabou
- Novartis Investigative Site, Abidjan, Côte d’Ivoire
- Novartis Investigative Site, Commune de La Kenya Lubumbashi, Du Haut Katanga, Democratic Republic of the Congo
- Novartis Investigative Site, Lambaréné, Gabon
- Mali (2):
  - Novartis Investigative Site, Kati
  - Novartis Investigative Site, Sotouba

IPD SHARING:
Plan to Share IPD: Yes
Novartis is commited to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Ogutu B, Yeka A, Kusemererwa S, Thompson R, Tinto H, Toure AO, Uthaisin C, Verma A, Kibuuka A, Lingani M, Lourenco C, Mombo-Ngoma G, Nduba V, N'Guessan TL, Nassa GJW, Nyantaro M, Tina LO, Singh PK, El Gaaloul M, Marrast AC, Chikoto H, Csermak K, Demin I, Mehta D, Pathan R, Risterucci C, Su G, Winnips C, Kaguthi G, Fofana B, Grobusch MP. Ganaplacide (KAF156) plus lumefantrine solid dispersion formulation combination for uncomplicated Plasmodium falciparum malaria: an open-label, multicentre, parallel-group, randomised, controlled, phase 2 trial. Lancet Infect Dis. 2023 Sep;23(9):1051-1061. doi: 10.1016/S1473-3099(23)00209-8. Epub 2023 Jun 13. PMID 37327809